CLINICAL TRIAL: NCT00612053
Title: Italian Registry on Treatment for Unprotected Left Main Disease (Registro Italiano Sul Trattamento Del Tronco coMune Non protettO)
Brief Title: Italian Registry on Unprotected Left Main
Acronym: RITMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Giuseppe Biondi Zoccai, Assistant Professor in Cardiology, University of Turin
Other Study IDs: CEI/167
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-02

CONDITIONS: Cardiovascular Disease; Coronary Artery Disease
Keywords: cardiovascular disease; coronary artery bypass grafting (CABG); coronary artery disease (CAD); percutaneous transluminal coronary angioplasty (PCI); unprotected left main disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The RITMO (Registro Italiano sul trattamento del Tronco coMune non protettO) observational study will appraise the prevalence, management strategy, and prognosis of unprotected left main coronary artery disease in Italy.

DETAILED DESCRIPTION:
The RITMO (Registro Italiano sul trattamento del Tronco coMune non protettO) observational study will be a prospective, multicenter, observational study aiming to appraise the prevalence, management strategy, and prognosis (up to 5 years) of unprotected left main coronary artery disease in Italy. A total of 45 Italian secondary and tertiary care centers will participate, and enroll patients during a period of 12 to 18 months. Patients will be included provided that they complete a written informed consent form and significant unprotected left main coronary artery disease is established at diagnostic coronary angiography. The primary end-point will be the 12-month rate of major adverse cerebro-cardiovascular events (ie death, myocardial infarction, stroke, or coronary revascularization).

ELIGIBILITY:
Inclusion Criteria:

* angiographic evidence of significant unprotected left main disease
* lack of patent bypass grafts for the left coronary system
* willingness to complete written informed consent form
* willingness to comply with subsequent follow-up contacts

Exclusion Criteria:

* lack of written informed consent form
* inability to comply with subsequent follow-up contacts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected coronary artery disease undergoing diagnostic coronary angiography.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
major adverse cerebro-cardiovascular events (ie death, myocardial infarction, stroke, or coronary revascularization) | 12 months

SECONDARY OUTCOMES:
major adverse cerebro-cardiovascular events | 60 months
Canadian Cardiac Society functional class | 60 months
quality of life (EuroQoL) | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Biondi Zoccai, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Division of Cardiology, University of Turin, Turin, To, Italy